CLINICAL TRIAL: NCT06036602
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Trial to Evaluate Safety, Tolerability, and Immune Responses of an Investigational Monovalent Chimpanzee Adenoviral-Vectored Sudan Ebolavirus Vaccine in Healthy Adults
Brief Title: Monovalent Chimpanzee Adenoviral-Vectored Sudan Ebolavirus Vaccine in Healthy Adults
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sabin-003
Record Dates: First submitted 2023-08-21; First posted 2023-09-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-01

CONDITIONS: Ebola Sudan Virus Disease
Keywords: Sudan Ebolavirus (SUDV); Sudan Ebolavirus Vaccine; cAD3-Ebolavirus Vaccine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 4:1 to receive the cAd3-Sudan Ebolavirus vaccine at 1.0 × 10^11 PU dose or placebo at Day 1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- cAD3-Sudan Ebolavirus Vaccine (Experimental): Single dose of cAd3-Sudan Ebolavirus vaccine (1x10^11 PU) administered intramuscularly (IM) with needle and syringe.
  Interventions: Biological: cAD3-Sudan Ebolavirus Vaccine
- Placebo (Placebo Comparator): 0.9% NaCl solution for injection)administered intramuscularly (IM) with needle and syringe in a volume of 0.56 mL
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: cAD3-Sudan Ebolavirus Vaccine — The recombinant chimpanzee adenovirus Type 3-vectored Sudan Ebolavirus vaccine, (cAd3-EBO S) is composed of a cAd3 vector that expresses wild type glycoprotein (WT GP) from the Sudan Gulu ebolavirus strain.
  Arms: cAD3-Sudan Ebolavirus Vaccine
Other: Placebo — 0.9% NaCl solution for injection.
  Arms: Placebo

SUMMARY:
A Phase 2, Randomized, Double-blind, Placebo-Controlled Trial to Evaluate Safety, Tolerability, and Immune Responses of an Investigational Monovalent Chimpanzee Adenoviral-Vectored Sudan Ebolavirus Vaccine in Healthy Adults

DETAILED DESCRIPTION:
This is a multi-center, double-blinded, placebo-controlled, Phase II study to evaluate safety, tolerability, and immunogenicity of a single dose of cAd3-Sudan Ebolavirus vaccine in healthy adults up to 70 years of age, in Uganda and Kenya. The study will enroll 125 eligible participants randomized 4:1 to receive the cAd3-Sudan Ebolavirus vaccine at 1.0 × 10^11 PU dose or placebo (0.9% sodium chloride (NaCl) solution) at Day 1, intramuscularly in deltoid muscle. Participants will be screened for eligibility up to 28 days before enrollment. Enrollment will be staggered, starting with healthy adults 18 to 50 years of age (inclusive). Upon enrollment of minimum 25 younger adult participants (sentinel), the safety data up to 7 days post vaccination of these 25 sentinel participants will be reviewed by the independent Data Safety Monitoring Board (DSMB). Progression to enrollment of the older adults (>50 to 70 years of age) will be dependent on the unblinded review of the DSMB. Safety and immunogenicity will be assessed at Days 1, 8, 15, 29, 85, 169, and will conclude at the end of study visit on Day 366.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete and provide written informed consent prior to any study procedure; including injection site photograph consent, completing an Assessment of Understanding (AoU) prior to enrollment by answering 9 out of 10 questions correctly at least once in 3 attempts, and including optional consent for retention of blood samples for potential future testing and assay development. Note: Participants can be enrolled even if they do not provide optional consent for retention of blood samples for potential future testing and assay development.
2. Able to read and write the language used in diary card.
3. Male or non-pregnant female 18 to 70 years of age (inclusive) at time of informed consent.
4. Is capable of understanding and agrees to comply with planned study procedures and to be available for all clinic follow-up for all planned study visits.
5. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
6. Has a means to be contacted and to contact the investigator during the study.
7. Agree not to receive any vaccine within 28 days from study vaccination (prior and after), with the exception of an emergency use authorization or authorized non-adenoviral vectored COVID-19 vaccine, which may be given within 14 days of study vaccination.
8. Agree not to donate bone marrow, blood, or blood products until 3 months after the study vaccination.
9. In good general health without clinically significant medical conditions, based on medical history, physical examination, vital signs, and clinical laboratory results as deemed acceptable by the principal investigator.
10. Clinical laboratory results within 28 days prior to vaccination within the site's laboratory reference ranges (or deemed not clinically significant by the principal investigator) for the following parameters: hematology (CBC including hemoglobin, WBC, RBC, total lymphocyte count); coagulation tests (prothrombin time, INR, fibrinogen); chemistry (C-reactive protein, d-dimer, ALT, AST, and serum creatinine). A laboratory result that is outside the reference range and is deemed not clinically significant by the principal investigator will not exclude the participant.
11. Has a BMI >17 and ≤37 at screening.

    Female participant-specific criteria:
12. Negative pregnancy serum test at screening, and negative urine pregnancy test before vaccination, if of reproductive potential.
13. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 24 weeks after study vaccination if assessed to be woman of childbearing potential UNLESS they fulfill one of the following criteria:

    * At least 1 year postmenopausal.
    * Surgically sterile.

    Male participants must agree:
14. Not to father a child or donate sperm through study end.
15. To use a barrier (condom) means of birth control from vaccination through study end, if assessed to be of reproductive potential.

Exclusion Criteria:

1. Pregnant or lactating female or plans to become pregnant or breastfeed starting from study vaccination through to study end.
2. Has any medical disease or condition that, in the opinion of the investigator, precludes study participation. This includes any acute, subacute, intermittent, or chronic medical disease or condition that:

   * would place the participant at an unacceptable risk of injury,
   * render the participant unable to comply with the requirements of the protocol,
   * or may interfere with the evaluation of responses or the participant's successful completion of the trial (chronic conditions that are well-controlled and medically stable, i.e., no change in treatment for medical reasons occurred in the last 6 months and are allowed at the discretion of the principal investigator, e.g., hypertension, asthma, thyroid disease). The medical disease or condition also includes any confirmed or suspected immunosuppressive or immunodeficient conditions resulting from disease (e.g., malignancy, HIV infection) or immunosuppressive/cytotoxic therapies (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
3. Serology screen positive for infectious diseases (hepatitis B, hepatitis C, HIV 1 and 2, syphilis).
4. Known history of prior exposure to SUDV or prior diagnosis of SUVD.
5. Current diagnosis of COVID-19 by Reverse Transcription Polymerase Chain Reaction (RT-PCR) or antigenic testing or current signs and symptoms of COVID-19. Participants may be enrolled 14 days post resolution of all signs and symptoms of COVID-19 or of testing positive for COVID-19 in asymptomatic participants.
6. History of or active status of any of the following clinically significant conditions:

   * Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
   * Allergic reaction to excipients in the study vaccine including gentamycin, neomycin or streptomycin or any other aminoglycoside.
   * Diabetes mellitus type 1 or type 2.
   * Active tuberculosis.
   * Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
   * Idiopathic urticaria within the last year.
   * Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), use of anticoagulant medications such as warfarin, apixaban, or dabigatran, or significant bruising or bleeding difficulties with IM injections or blood draws.
   * Major thrombotic event or heparin-induced thrombocytopenia or Vaccine-Induced Thrombotic Thrombocytopenia (VITT).
   * Malignancy of any organ system, treated or untreated, within the past 5 years from screening (if diagnosed malignancy is 5 or more years prior to enrollment and cured with no ongoing treatment it will NOT be considered an exclusion).
   * Seizure in the past 3 years or treatment for seizure disorder in the past 3 years.
   * Asplenia or functional asplenia.
   * Autoimmune disease/autoinflammatory condition.
   * Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent.
7. Has a clinically significant acute illness (this does not include minor illnesses) or temperature ≥38.0°Celsius (≥100.4° Fahrenheit) within 24 hours of the planned dose of study vaccine. Re-evaluation of eligibility may be performed at resolution of all signs and symptoms, and randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor (as appropriate).
8. Receipt of any of the following substances:

   * COVID-19 vaccine that has not received emergency use authorization or approval per local regulatory agency.
   * Prior receipt of Ebola or Marburg vaccine.
   * Prior receipt of any adenoviral-vectored vaccine, adenovirus-based or adeno-associated virus (AAV)-based gene therapies or treatments, including adenoviral COVID-19 vaccines or boosters.
   * Participant received an investigational drug (including investigational drugs for prophylaxis of COVID-19) within 28 days of dosing or within washout period (5 half-lives) of such drug or has used an invasive investigational medical device within 28 days of dosing.
   * Received investigational Ig or monoclonal antibodies within 3 months.
   * Received convalescent serum for COVID-19 treatment within 3 months.
   * Received an investigational vaccine within 3 months before the planned administration of the first dose of study vaccine.
   * Is currently enrolled or plans to participate in another investigational or interventional study during this study (observational/registry studies are allowed).
9. Use of immunomodulators or systemic glucocorticoids in daily doses of glucocorticoid equivalence >20 mg of prednisolone in the last 90 days, and for periods exceeding 10 days. Non-Steroidal Anti-Inflammatory Drugs (NSAIDS) are permitted.
10. Receipt of blood products within 3 months prior to enrollment.
11. Current anti-tuberculosis prophylaxis or therapy.
12. Abnormality or permanent body art (such as tattoo) in deltoid region that would interfere with ability to observe or assess injection site reactions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of cAd3-Sudan Ebolavirus vaccine through the assessment of SAEs, solicited AEs, unsolicited AEs, AESI, MAAE, and AE | 1 year
  Count and percentage of vaccinated participants who develop:
  * serious adverse events (SAEs),
  * solicited adverse events (AEs),
  * unsolicited AEs,
  * adverse event of special interest (AESI),
  * medically attended adverse events (MAAE),
  * AE at each intensity level.
  Estimand 1a (Primary): Count and percentage of vaccinated participants who would develop SAEs, solicited AEs, unsolicited AEs, AESI, MAAE, and AE at each intensity level will be evaluated with each treatment group. A treatment policy strategy is used for assessing safety irrespective of a current (or prior) infection at time of the vaccination. Infections and death (if they meet the AE and time window criteria) are included in the endpoint (composite strategy).

SECONDARY OUTCOMES:
To evaluate the antibody response (IgG) to cAd3-EBO S vaccine at Day 29 post-vaccination. | 1 month
  Secondary Endpoint: GMC of anti-Sudan Ebolavirus-GP binding IgG antibodies at Day 29 post-vaccination. Estimand 2a: geometric mean concentration (GMC) of the vaccine group will be compared to placebo at Day 29 post-vaccination. The hypothetical strategy is used to estimate antibody levels without subsequent Sudan Ebolavirus (SUDV) infection or influence from immune-modifying drugs or non-study vaccines. The principal stratum strategy excludes those with active or prior SUDV infection at the time of the vaccination.

CONTACTS AND LOCATIONS:
Locations (2):
- KEMRI/Centre for Respiratory Disease Research Siaya Clinical Research Annex, Siaya, Kenya
- Makerere University-Walter Reed Project, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The clinic trial results will be published in a peer-reviewed journal, which will include, as feasible, the study protocol. A summary of the study results will be included within the trial registration records in ClinicalTrials.gov.
Supporting Information: Study Protocol